CLINICAL TRIAL: NCT03396432
Title: The Videolaryngoscopy in Small Infants (VISI) Trial
Brief Title: The Videolaryngoscopy in Small Infants
Acronym: VISI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-014302
Record Dates: First submitted 2017-12-19; First posted 2018-01-11 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Surgery; Anesthesia, Endotracheal
Keywords: laryngoscope; intubation; first attempt success; oxygen saturation; airway management; Videolaryngoscopy; Direct laryngoscopy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multi-center parallel group trial
Who Masked: Outcomes Assessor
Masking Description: Statistician will be blinded at the time of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Video Laryngoscopy for endotracheal (ET) Placement (Active Comparator): Device:
  Storz C-MAC Video Laryngoscope
  Interventions: Device: Video Laryngoscopy for ET placement; Device: Direct Laryngoscopy for ET Placement
- Direct Laryngoscopy for ET Placement (Active Comparator): Device:
  Miller Laryngoscope
  Interventions: Device: Video Laryngoscopy for ET placement; Device: Direct Laryngoscopy for ET Placement

INTERVENTIONS:
Device: Video Laryngoscopy for ET placement — Tracheal intubation performed with the Storz C-Mac Video Laryngoscope
Device: Direct Laryngoscopy for ET Placement — Tracheal Intubation performed with the Miller Blade

SUMMARY:
Complications related to infant (≤ 1 year) airway management are under-appreciated because of few rigorous and targeted studies. Investigators have recently shown that multiple tracheal intubation (TI) attempts are a key risk factor for intubation-related complications in small children. Tracheal Intubation using Video laryngoscopy (VL) has become popular in anesthesiology practice because of several advantages over conventional direct laryngoscopy (DL). Studies show that VL improves the view of the airway compared to DL, requires fewer intubation attempts, but may take more time to intubate the trachea. This study compares first attempt success of VL to DL in infants presenting for elective surgery.

DETAILED DESCRIPTION:
Objectives:

* Primary Objective To compare the tracheal intubation (TI) first attempt success rate using VL vs. DL in children ≤ 12 months old.
* Secondary Objectives To compare the lowest oxygen saturation during tracheal intubation with VL vs. DL.

Study Design:

Prospective, randomized, multi-center parallel group trial

Setting/Participants:

This will be a multi-center study with a minimum of four participating centers. The target population will be children ≤ 12 months age scheduled for elective surgery requiring general anesthesia with endotracheal intubation.

Study Interventions and Measures:

The study intervention will be a 1:1 randomization to perform tracheal intubation with the Storz C-Mac Miller 1 (VL) or the conventional Miller laryngoscope (DL).

Main study outcome measures are as follows:

* The first intubation attempt success rate with each device
* The number of attempts for successful intubation with each device
* Complications associated with intubation

ELIGIBILITY:
Inclusion Criteria

1. Males or females age 0 to <12 months.
2. Scheduled for non-cardiac surgery or procedure lasting longer than 30 minutes under general anesthesia where oral endotracheal intubation will be performed by an anesthesiology clinician.
3. Subject/Parental/guardian permission (informed consent).

Inclusion for clinician participants:

1) Pediatric anesthesia attending, pediatric anesthesia fellows, and anesthesia resident

Exclusion Criteria

1. History of difficult intubation
2. History with abnormal airway
3. Predictive of difficult intubation upon physical examination
4. Parents/guardians who, in the opinion of the investigator, may be unable to understand or give informed consent

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 566 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fiadjoe, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Princess Margaret Hospital For Children, Subiaco, Perth, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Sun H, Liu M, Lin Z, Jiang H, Niu Y, Wang H, Chen S. Comprehensive identification of 125 multifarious constituents in Shuang-huang-lian powder injection by HPLC-DAD-ESI-IT-TOF-MS. J Pharm Biomed Anal. 2015 Nov 10;115:86-106. doi: 10.1016/j.jpba.2015.06.013. Epub 2015 Jun 30. PMID 26177215
- [Background] Lingappan K, Arnold JL, Shaw TL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2015 Feb 18;(2):CD009975. doi: 10.1002/14651858.CD009975.pub2. PMID 25691129
- [Background] Goto T, Gibo K, Hagiwara Y, Morita H, Brown DF, Brown CA 3rd, Hasegawa K; Japanese Emergency Medicine Network Investigators. Multiple failed intubation attempts are associated with decreased success rates on the first rescue intubation in the emergency department: a retrospective analysis of multicentre observational data. Scand J Trauma Resusc Emerg Med. 2015 Jan 16;23:5. doi: 10.1186/s13049-014-0085-8. PMID 25700237
- [Background] Goto T, Watase H, Morita H, Nagai H, Brown CA 3rd, Brown DF, Hasegawa K; Japanese Emergency Medicine Network Investigators. Repeated attempts at tracheal intubation by a single intubator associated with decreased success rates in emergency departments: an analysis of a multicentre prospective observational study. Emerg Med J. 2015 Oct;32(10):781-6. doi: 10.1136/emermed-2013-203473. Epub 2014 Dec 31. PMID 25552546
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Souza Nd, Carvalho WB. [Complications of tracheal intubation in pediatrics]. Rev Assoc Med Bras (1992). 2009 Nov-Dec;55(6):646-50. Portuguese. PMID 20191217
- [Background] Grunwell JR, Kamat PP, Miksa M, Krishna A, Walson K, Simon D, Krawiec C, Breuer R, Lee JH, Gradidge E, Tarquinio K, Shenoi A, Shults J, Nadkarni V, Nishisaki A; National Emergency Airway Registry for Children (NEAR4KIDS) and the Pediatric Acute Lung Injury and Sepsis (PALISI) Network. Trend and Outcomes of Video Laryngoscope Use Across PICUs. Pediatr Crit Care Med. 2017 Aug;18(8):741-749. doi: 10.1097/PCC.0000000000001175. PMID 28492404
- [Background] Abdelgadir IS, Phillips RS, Singh D, Moncreiff MP, Lumsden JL. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in children (excluding neonates). Cochrane Database Syst Rev. 2017 May 24;5(5):CD011413. doi: 10.1002/14651858.CD011413.pub2. PMID 28539007
- [Background] Nouruzi-Sedeh P, Schumann M, Groeben H. Laryngoscopy via Macintosh blade versus GlideScope: success rate and time for endotracheal intubation in untrained medical personnel. Anesthesiology. 2009 Jan;110(1):32-7. doi: 10.1097/ALN.0b013e318190b6a7. PMID 19104167
- [Background] Howard-Quijano KJ, Huang YM, Matevosian R, Kaplan MB, Steadman RH. Video-assisted instruction improves the success rate for tracheal intubation by novices. Br J Anaesth. 2008 Oct;101(4):568-72. doi: 10.1093/bja/aen211. Epub 2008 Aug 1. PMID 18676418
- [Derived] Garcia-Marcinkiewicz AG, Kovatsis PG, Hunyady AI, Olomu PN, Zhang B, Sathyamoorthy M, Gonzalez A, Kanmanthreddy S, Galvez JA, Franz AM, Peyton J, Park R, Kiss EE, Sommerfield D, Griffis H, Nishisaki A, von Ungern-Sternberg BS, Nadkarni VM, McGowan FX Jr, Fiadjoe JE; PeDI Collaborative investigators. First-attempt success rate of video laryngoscopy in small infants (VISI): a multicentre, randomised controlled trial. Lancet. 2020 Dec 12;396(10266):1905-1913. doi: 10.1016/S0140-6736(20)32532-0. PMID 33308472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was recruited per protocol without any protocol deviation or violation.
Pre-assignment Details: The block size was varying among 2, 4, 6 to avoid the predictability of device assignment. To further balance device assignment, we'll stratify the randomization by study site and clinician's role. Separate randomization schedule was generated for each stratum.
Groups:
- Video Laryngoscopy for Endotracheal (ET) Placement: Device:
  Storz C-MAC Video Laryngoscope
  Video Laryngoscopy for ET placement: Tracheal intubation performed with the Storz C-Mac Video Laryngoscope
  Direct Laryngoscopy for ET Placement: Tracheal Intubation performed with the Miller Blade
- Direct Laryngoscopy for ET Placement: Device:
  Miller Laryngoscope
  Video Laryngoscopy for ET placement: Tracheal intubation performed with the Storz C-Mac Video Laryngoscope
  Direct Laryngoscopy for ET Placement: Tracheal Intubation performed with the Miller Blade
Period: Overall Study
Arm/Group | Video Laryngoscopy for Endotracheal (ET) Placement | Direct Laryngoscopy for ET Placement
Started | 283 | 283
Completed | 274 | 277
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Population: 566 subjects enrolled with 551 evaluable
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Laryngoscopy for Endotracheal (ET) Placement | Direct Laryngoscopy for ET Placement | Total
Number analyzed (Participants) | 274 | 277 | 551
Age, Customized [Count of Participants; unit: Participants]
  0-30 Days | 17 | 20 | 37
  31-90 Days | 55 | 64 | 119
  > 90 Days | 202 | 193 | 395
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 96 | 175
  Male | 195 | 181 | 376
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 6.5 [4.64 to 8.18] | 6.6 [4.89 to 8.34] | 6.5 [4.74 to 8.26]
ASA [Count of Participants; unit: Participants]
  1 - Normal | 58 | 72 | 130
  2 - Mild systemic disease | 133 | 136 | 269
  >= 2 - Mod - Severe systemic disease | 83 | 69 | 152
Induction Technique -IV [Count of Participants; unit: Participants] | 28 | 39 | 67
Muscle Relaxant [Count of Participants; unit: Participants]
  None | 15 | 14 | 29
  Succinylcholine | 9 | 11 | 20
  Other | 250 | 252 | 502
Device experience as number of infant intubations [Count of Participants; unit: Participants]
  0 | 38 | 10 | 48
  1-10 | 79 | 59 | 138
  11-20 | 36 | 36 | 72
  21-50 | 49 | 37 | 86
  >50 | 62 | 128 | 190
  Unknown | 10 | 7 | 17
Provider Role [Count of Participants; unit: Participants]
  Anes Attending | 69 | 69 | 138
  Anes Fellow | 99 | 102 | 201
  Anes Resident | 106 | 106 | 212

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Success in the First Attempt
Description: comparing the tracheal intubation (TI) first attempt success rate using VL vs. DL
Time Frame: at the time of intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscopy for Endotracheal (ET) Placement | Direct Laryngoscopy for ET Placement
Number analyzed (Participants) | 274 | 277
Participants | 253 | 243

2. Secondary Outcome: Hypoxia
Description: Comparing the lowest oxygen saturation during tracheal intubation with VL vs. DL
Time Frame: At the time of intubation
Measure: Count of Participants; unit: Participants
Groups:
- Video Laryngoscopy for Endotracheal (ET) Placement: Device:
  Storz C-MAC Video Laryngoscope
  Video Laryngoscopy for ET placement: Tracheal intubation performed with the Storz C-Mac Video Laryngoscope
- Direct Laryngoscopy for ET Placement: Device:
  Miller Laryngoscope
  Direct Laryngoscopy for ET Placement: Tracheal Intubation performed with the Miller Blade
Arm/Group | Video Laryngoscopy for Endotracheal (ET) Placement | Direct Laryngoscopy for ET Placement
Number analyzed (Participants) | 274 | 277
Participants | 9 | 15

ADVERSE EVENTS:
Time Frame: Upon discharge from PACU or up to 24 hr after intubation
Arm/Group | Video Laryngoscopy for Endotracheal (ET) Placement | Direct Laryngoscopy for ET Placement
All-Cause Mortality (participants affected / at risk) | 0/274 | 0/277
Serious Adverse Events (participants affected / at risk) | 0/274 | 0/277
Other Adverse Events (participants affected / at risk) | 3/274 | 2/277
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video Laryngoscopy for Endotracheal (ET) Placement (N=274) | Direct Laryngoscopy for ET Placement (N=277)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cleft palate repair-Possibly related
Intermittent tachypnea (Cardiac disorders) | 1 (1) | 0 (0) — History of respiratory failure-Not related
Brief Desaturation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) — Probably not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT03396432/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT03396432/ICF_001.pdf